CLINICAL TRIAL: NCT04895657
Title: Extended-infusion Piperacillin-Tazobactam Versus Intermittent-Infusion Dosing Strategy in Critically Ill Patients With Suspected or Confirmed Bacterial Infections.
Brief Title: Extended-infusion of Piperacillin-Tazobactam Versus Intermittent Infusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Christina Medhat, Teaching assistant, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 198
Record Dates: First submitted 2021-04-19; First posted 2021-05-20 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Gram-Negative Infections
Keywords: Antibiotics; Beta-lactams; Continuous administration
MeSH Terms: interventions — Piperacillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Piperacillin/Tazobactam Intermittent infusion (Other): 4.5 gm Piperacillin/Tazobactam I.V intermittent over 30 min. every 8 hours.
  Interventions: Drug: Piperacillin/Tazobactam Intermittent infusion
- Piperacillin/Tazobactam Continuous infusion (Other): 4.5 gm Piperacillin/Tazobactam I.V extended infusion over 4 hours every 8 hours.
  Interventions: Drug: Piperacillin/Tazobactam Continuous infusion

INTERVENTIONS:
Drug: Piperacillin/Tazobactam Continuous infusion — Continuous infusion
  Other Names: Piprataz injection
  Arms: Piperacillin/Tazobactam Continuous infusion
Drug: Piperacillin/Tazobactam Intermittent infusion — Intermittent infusion
  Other Names: Piprataz injection
  Arms: Piperacillin/Tazobactam Intermittent infusion

SUMMARY:
Continuous-infusion of piperacillin/tazobactam over 4 hrs instead of 30-minute intermittent dosage regimen has shown observable outcomes. Our objective is to assess whether continuous infusion of piperacillin/tazobactam is superior in terms of efficacy, safety and cost to the intermittent regimen to treat suspected or proved infections due to gram negative bacteria. The setting is Critical Care Medicine Department at Cairo University Hospitals. Methods A prospective randomized comparative study.

DETAILED DESCRIPTION:
A total of 56 patients were recruited from ICU- Cairo University Hospitals. All adult critically ill patients admitted to Critical Care Medicine Department with suspected or confirmed bacterial infections on admission or during their ICU stay were assessed for inclusion into the study. All patients were subjected to the following: A. Patient's full history: Age, sex ,medical history ,concurrent diseases, concurrent medications

B. Patient evaluation and assessment:

The following were evaluated at baseline and periodically thereafter until day of stopping antibiotic, discharge and/or death :

1. Kidney functions (Serum creatinine, blood urea nitrogen)
2. Liver functions (ALT, AST, Bil D, Bil T, Albumin)
3. Complete blood count
4. Microbiological Evaluation: Cultures and sensitivity tests from suspected site of infection
5. Clinical signs and symptoms of infection documented by the attending physician on patient's medical record
6. APACHE II Variables

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-74 years
* Expected ICU stay more than 24 hours

Exclusion Criteria:

* Allergy or potential allergy to the study medications

  * Pregnancy
  * Patients with CrCl< 20 ml/min or on dialysis
  * Cancer patients

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2020-01-26 (Actual); Study Completion 2020-01-26 (Actual)

PRIMARY OUTCOMES:
Clinical cure | ICU length of stay, assessed up to 30 days
  Clinical cure, expressed in percentage, will be considered fulfilled if all the following criteria are met : Cure or improvement of clinical signs and symptoms caused by the infection, normalized WBCs and body temperature.
Total cost | ICU length of stay, assessed up to 30 days
  Cost in Dollars (prices of drugs ,supplies prices, preparation, administration, daily hospital stay cost )

SECONDARY OUTCOMES:
ICU Length of stay | ICU length of stay, assessed up to 30 days
  ICU Length of stay in Days
Mortality | ICU length of stay, assessed up to 30 days
  percentage
Readmission within 30- days | 30 days
  Days
Adverse drug events | ICU length of stay, assessed up to 30 days
  Any adverse event occurring during study drug administration

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/57/NCT04895657/Prot_SAP_000.pdf